CLINICAL TRIAL: NCT07258485
Title: A Study to Evaluate Sleep Electroencephalogram (EEG) Features in Participants With Major Depressive Disorder (MDD)
Brief Title: A Study to Evaluate Sleep Electroencephalogram (EEG) Features (Brain Activity While Sleeping) in Participants With Major Depressive Disorder (MDD)
Status: Recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 42847922MDD3014; 42847922MDD3014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants With Major Depressive Disorder with Moderate to Severe Insomnia Symptoms (MDDIS): The MDDIS cohort includes participants with moderate to severe insomnia symptom severity as measured by clinical outcome assessments during the screening phase.
- Participants With MDD With No Or Mild Insomnia Symptoms (Non-MDDIS): The Non-MDDIS cohort includes participants with no or mild insomnia symptoms as measured by clinical outcome assessments during the screening phase.

SUMMARY:
The purpose of this study is to evaluate sleep in participants with Major Depressive Disorder with moderate to severe insomnia symptoms (MDDIS) or MDD with no or mild insomnia symptoms (non-MDDIS), using an at-home sleep Electroencephalogram (EEG; a device that records brain activity during sleep). The study also aims to examine the association between objective sleep EEG features (measured using devices) and subjective sleep measures (self-reported experiences, such as how a person feels about their sleep) in participants with MDDIS or non-MDDIS.

ELIGIBILITY:
Inclusion criteria:

* Participants must be medically stable, based on investigator review of medical history, vital signs (including blood pressure), and clinical judgment. In cases of any medical concern, the investigator has the option to perform local 12-lead electrocardiogram (ECG) or local clinical laboratory testing at screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* Meet diagnostic and statistical manual of mental disorders (5th edition) (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 axis I disorders-clinical trials version (SCID-CT). Must be diagnosed with first depressive episode prior to age 60
* Have had an inadequate response to at least 1 but no more than 2 antidepressants, administered at an adequate dose and duration started in the current episode of depression. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression. An inadequate response is defined as less than (<) 50 percent (%) reduction but with some improvement (that is, improvement greater than [>] 0%) in depressive symptom severity with residual symptoms present, and overall good tolerability, as assessed by the massachusetts general hospital-antidepressant treatment response questionnaire (MGH-ATRQ). An adequate trial is defined as an antidepressant treatment for at least 6 weeks on a stable dose at or above the minimum therapeutic dose specified in the MGH-ATRQ, and this must include the participant's current antidepressant treatment
* Is receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any formulation and approved by the Food and Drug Administration (FDA): citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at therapeutic dose level per MGH-ATRQ) for at least 6 weeks
* Has a body mass index (BMI) of 18 to 40 kilograms per meter square (Kg/m^2), inclusive

Exclusion criteria:

* Had major surgery (for example, requiring general anesthesia) within 2 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Has a history of treatment-resistant MDD, defined as a lack of response to 2 or more adequate antidepressant treatments in the current episode, as indicated by no or minimal (less than or equal to [<=] 25%) improvement in symptoms when treated with an antidepressant of adequate dose (per MGH-ATRQ) and duration (at least 6 weeks)
* Has a primary DSM-5 diagnosis of panic disorder, generalized anxiety disorder, social anxiety disorder, or specific phobia which has been the primary focus of psychiatric treatment within the past 2 years. These are allowed as secondary diagnoses if MDD is the primary focus of treatment according to the investigator
* Has a history or current diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, or somatoform disorders
* Has cognitive impairment per investigator judgment that would render the informed consent invalid or limit the ability of the participant to comply with the study requirements. Participant has neurodegenerative disorder (for example, alzheimer's disease, vascular dementia, parkinson's disease with clinical evidence of cognitive impairment) or evidence of mild cognitive impairment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with MDD with moderate to severe insomnia symptoms (MDDIS) or MDD with no or mild insomnia symptoms (non-MDDIS).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Characterization of Objective Sleep Electroencephalogram (EEG) Features in Major Depressive Disorder Participants with Moderate to Severe Insomnia Symptoms (MDDIS) or Non-MDDIS As Assessed by Dreem 3S Headband | Day -7 to Day -1
  Objective sleep EEG features in MDD participants will be assessed using dreem 3S headband. It will be used in this study to capture macro and micro sleep architecture including sleep initiation (latent to persistent sleep, sleep onset latency), sleep maintenance (rapid eye movement [REM] latency, total sleep time, REM percentage, and duration) and arousal features (stage shift index, number of awakenings). It also uses a 3D accelerometer to measure movements, head position, and respiratory rate/trace during sleep.
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by Consensus Sleep Diary (CSD) | Day -6 to Day 1
  Subjective sleep EEG features in MDD participants will be assessed using CSD. Participants will be asked to provide answers to questions to determine their subjective experience of nighttime sleep, daytime napping/dozing, feeling refreshed upon awakening, and the usage of over-the-counter and prescription sleep aids and the Dreem 3S headband by recording their answers in a daily sleep diary (CSD). CSD will be used in this study to capture the parameters including self-reported sleep onset latency, subjective total sleep time, subjective wake after sleep onset, subjective number of nighttime awakenings, subjective quality of sleep, subjective refreshed feeling on waking, self-reported number of naps, self-reported nap time, self-reported sleep aids, self-reported sleep impact while utilizing Dreem 3S headband.
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by the Structured Interview Guide (SIGH-D) Used to Implement the 17 item Hamilton Depression Rating Scale (HRSD17) | Day -7 to Day -1
  Subjective sleep EEG features in MDD participants will be assessed using SIGH-D used to implement HRSD17 scale. The structured interview guide SIGH-D will be used to implement the HRSD17. HRSD17 scale contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a Likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-54.
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD)- 8a Short Forms | Day -7 to Day -1
  Subjective sleep EEG features in MDD participants will be assessed using PROMIS-SD-8a. PROMIS-SD-8a uses all items on the 8a form. The PROMIS-SD instrument assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Sleep Disturbance does not focus on symptoms of specific sleep disorders, nor does it provide subjective estimates of sleep quantities (total amount of sleep, time to fall asleep, amount of wakefulness during sleep).
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by PROMIS-SD- 4a Short Forms | Day -7 to Day -1
  Subjective sleep EEG features in MDD participants will be assessed using PROMIS-SD-4a. PROMIS-SD-4a uses 4 of the 8 items on the 8a form. The PROMIS-SD instrument assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Sleep Disturbance does not focus on symptoms of specific sleep disorders, nor does it provide subjective estimates of sleep quantities (total amount of sleep, time to fall asleep, amount of wakefulness during sleep).
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by PROMIS-SD- 10a Short Forms | Day -7 to Day -1
  Subjective sleep EEG features in MDD participants will be assessed using PROMIS-SD-10a. PROMIS-SD-10a uses all items on both the 8a and 2a forms. The PROMIS-SD instrument assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Sleep Disturbance does not focus on symptoms of specific sleep disorders, nor does it provide subjective estimates of sleep quantities (total amount of sleep, time to fall asleep, amount of wakefulness during sleep).
Characterization of Subjective Sleep Measures in MDD Participants with MDDIS or Non-MDDIS As Assessed by Insomnia Severity Index (ISI) | Day -7 to Day -1
  Subjective sleep EEG features in MDD participants will be assessed using patient and clinician version of ISI. The clinician version of the ISI will be completed by an independent rater. The ISI is a 7-item questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance, early morning awakening problems; sleep dissatisfaction; interference of sleep problem with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale (0-4) is used to rate each item, yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0 7); sub threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Behavioral Research Specialists LLC, Glendale, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Velocity Clinical Research, Hallandale, Florida
  - Meridian International Research, Miami Gardens, Florida
  - Chicago Research Center, Chicago, Illinois
  - Adams Clinical, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Adams Clinical, New York, New York
  - Adams Clinical, The Bronx, New York
  - Adams Clinical, DeSoto, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency